CLINICAL TRIAL: NCT05707260
Title: Effectiveness of the CDK-SMS Nursing Intervention for Adults With Chronic Kidney Disease
Brief Title: Effectiveness of the CDK-SMS Intervention for Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Judith Medellin Olaya (Other)
Responsible Party: Sponsor-Investigator, Judith Medellin Olaya, Principal Investigator, Universidad Nacional de Colombia
Organization: Universidad Nacional de Colombia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 026-21
Record Dates: First submitted 2023-01-18; First posted 2023-01-31 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD SMS intervention (Active Comparator): CKD SMS (Chronic Kidney Disease Self-Management Support) intervention (6,27), guided by the Social Cognitive Theory, through the manipulation of self-efficacy, is educational for the adult with CKD in early stages where a primer will be used which contains a primer that explains the functions of the kidneys, the first signs and symptoms of CKD and the strategies to control or delay the progression of CKD, such as the benefits of maintaining a healthy lifestyle and adherence to treatment. Also, a diary for participants to record side effects of medications, monitor their clinical data, treatment plan and questions for medical appointments.
  Interventions: Behavioral: CKD SMS
- Conventional intervention (No Intervention): The conventional intervention corresponds to the protocol established in the program of the renal unit for the management of people with CKD in early stages.

INTERVENTIONS:
Behavioral: CKD SMS — The intervention begins with a face-to-face or digitally assisted session, entry into improving the knowledge and self-management of CKD through, using the four sources of manipulation of self-efficacy (achievement of performance, indirect experience, verbal persuasion, and self-evaluation). In this session, participants will be asked to identify their problems related to CKD and establish, based on these two goals, that they are real and achievable according to their priorities. These goals will be recorded in the monitoring format and will be monitored in the telephone or WhatsApp follow-ups. This using the performance achievement manipulation source, said session lasts 60 minutes, as does the final session at week 16.
  Arms: CKD SMS intervention

SUMMARY:
Type of Study: a pragmatic randomized clinical trial. Research question How effective is the CKD SMS self-management nursing intervention on self-management behaviors, self-efficacy, and adherence in adults with early-stage CKD compared to usual care? General objective To determine the effectiveness of the self-management nursing intervention (CKD SMS) on self-management behaviors, self-efficacy, and therapeutic adherence in people with CKD in early stages compared to usual care.

Target population: Adult men and women with chronic kidney disease in stages 1-4, with different characteristics such as educational level, socioeconomic status, and marital status. Taking into account that the definition of early stages through the criteria demarcated by the Colombian clinical practice guideline, where the glomerular filtration rate (GFR) is the indicator for stratification as follows: stage 1 people with a GFR less than or equal to 90 (ml (min / 1.73 m2), stage 2 people with GFR between 60-89 (ml (min / 1.73 m2), stage 3 people with GFR between 30-59 (ml (min / 1.73 m2)) and stage 4 people with GFR between 15-30 (ml (min / 1.73 m2) who attend kidney protection programs of the Renal Units in Colombia.

STUDY VARIABLES

Among the variables that are available for the present study are:

* Independent Variables: Sociodemographic characteristics, related to the disease or clinical condition and the CKD intervention.
* Dependent variables: Self-management behaviors, therapeutic adherence, and self-efficacy.

Within the mediating, shaping or confounding variables, the following are found according to what is established in the literature: age, gender, level of education, time of diagnosis and other comorbidities, which are initially considered independent variables and will be measured. In the study, for its management, strategies such as randomization will be used, the differences between the crude estimates of an association and those adjusted considering a confounding variable will be identified and its adjustment is responsible for at least 10% in the magnitude of the difference.

INTERVENTIONS

* CKD SMS intervention CKD SMS (Chronic Kidney Disease Self-Management Support) intervention
* Conventional intervention The conventional intervention corresponds to the protocol established in the program of the renal unit for the management of people with CKD in early stages.

DETAILED DESCRIPTION:
Scope and justification of the proposal

Chronic kidney disease is a complex pathology, where the person who suffers from it is faced with unexpected changes in their customs and lifestyles, in addition to complying with a strict therapeutic regimen, because from its diagnosis it seeks to delay the progress of this, and the prevention of complications derived from its development. Within the disease management guidelines at the European level, which were necessary for the Colombian context, they recommend that the factors associated with disease progression should be addressed, which include: "the cause of the disease, the level of the glomerular filtration rate, the level of albuminuria, age, sex, race/ethnicity, elevated blood pressure, hyperglycemia, dyslipidemia, smoking, obesity, history of cardiovascular disease, continued exposure to nephrotoxic agents and others", most of which are modifiable, through self-management interventions.

Self-management interventions aimed at adults with CKD in its early stages contribute to improving the quality of life, self-management behaviors, and self-efficacy, but above all in the prevention of complications derived from the disease. Preventing a person with CKD from progressing to advanced stages or terminal management phases leads to lower healthcare costs by delaying the start of specialized treatments (renal replacement therapies) that require high technology and preventing complications that can lead to increased mortality in the population. Results that have been considered within health policies and therefore have become a premise that justifies the relevance of the nursing intervention in self-management.

The nursing intervention in self-management implies advancing in approaches where adults with early-stage CKD are active agents in managing their own care towards awareness and responsibility for the daily care of the disease. Today there is a nursing intervention in self-management the CKD SMS, designed specifically for the population object of this study, which has been administered in two countries where there are different socio-economic and cultural characteristics (Vietnam and Australia), demonstrating feasibility in its implementation and acceptability by the participants, in addition to being effective in promoting self-management behaviors, a comprehensive and novel construct, which is achieved through the manipulation of self-efficacy.

In the present proposal, therapeutic adherence is a central concept since it is expected that when performing the nursing intervention in self-management, adherence to the therapeutic regimen will increase, evidenced in the exercise of healthy habits, such as the intake of a diet in accordance with its condition and the reduction of risk factors inherent to the disease, also translated into the impact of these factors on clinical control variables such as: improving blood pressure control, glycosylated hemoglobin levels, but also an important impact in delaying the progression of the disease, which is evidenced not only by not requiring renal replacement therapies, but also by maintaining or improving the glomerular filtration rate, which is beneficial for both the person and for the health system.

The nursing professional plays an important role in the execution of self-management interventions such as the CKD SMS, since it is who within the health team has the responsibility of imparting education and monitoring people, in the investigations found in most of the Regarding the interventions that have been carried out, the participation of the nursing professional has been fundamental since it is the one who is in constant interaction with the person.

RESEARCH QUESTION

How effective is the CKD SMS (Chronic Kidney Disease Self-Management Support) self-management nursing intervention on self-management behaviors, self-efficacy, and adherence in adults with early-stage CKD compared to usual care?

OBJECTIVES

General objective

To determine the effectiveness of the self-management nursing intervention (CKD SMS) on self-management behaviors, self-efficacy, and therapeutic adherence in people with CKD in early stages compared to usual care.

Specific objectives

1. Describe the sociodemographic and clinical characteristics of the control group and the experimental group.
2. Establish the level of self-efficacy, self-management behaviors and therapeutic adherence as a baseline in people with chronic kidney disease in early stages.
3. To evaluate the changes in self-management behaviors, self-efficacy, and therapeutic adherence post-intervention and in the control group at 16 weeks.

Methodology This is a quantitative investigation, with a pragmatic randomized clinical trial (pRCT) design, parallel experimental type, given the one-to-one allocation in two parallel groups with repeated pre-test and post-test measures, considering that this type of study it is useful for evaluating interventions in usual care. In CKD, the use of a pRCT enables a broader range of patients to be included to test an intervention applicable to patient care and to measure relevant patient-centered outcomes, thus improving external validity and translation of the results into the clinical care.

Where the outcome variables are: Self-management behaviors (primary), self-efficacy and therapeutic adherence (secondary). The population will be adult men and women with chronic kidney disease in stages 1-4, who attend control of their disease or belong to the program.

Target population: Adult men and women with chronic kidney disease in stages 1-4, with different characteristics such as educational level, socioeconomic status, and marital status. Taking into account that the definition of early stages through the criteria demarcated by the Colombian clinical practice guideline, where the glomerular filtration rate (GFR) is the indicator for stratification as follows: stage 1 people with a GFR less than or equal to 90 (ml (min / 1.73 m2), stage 2 people with GFR between 60-89 (ml (min / 1.73 m2), stage 3 people with GFR between 30-59 (ml (min / 1.73 m2)) and stage 4 people with GFR between 15-30 (ml (min / 1.73 m2) who attend kidney protection programs of the Renal Units in Colombia.

Accessible population: Adult population men and women with chronic kidney disease in stages 1-4, with different characteristics such as educational level, socioeconomic status, marital status, those who attend control of their disease or belong to the predialysis in Colombia, which can be found in the databases provided by Renal Unit.

SAMPLE Sample design: The sample size was calculated through probability sampling, since individuals have the same probability of being chosen. On the other hand, of the comparison of means in independent groups, assuming a power of 80%, a confidence level of 95%, an expected mean difference of 18.13 in the improvement of self-management, reported by previous studies.

Sample size: A total of 82 participants (41 per group), in addition, a mortality of 20% of the participants is expected, so a total sample of 100 participants (50 per group) will be assumed. made in the Epidat 3.1 program.

Randomization: Participants will be randomized into two groups, using sequentially numbered opaque sealed envelopes, where the investigator and participants will be blinded to the allocation of each group. For the generation of the randomization sequence, it will be developed by the investigator by means of the realization of a table of random numbers in the Epidat 3.1 program to eliminate the selection bias, in the same way, said table will be verified to guarantee balance between the number of participants assigned to each group (control and intervention).

Blinding: In view of the need to minimize bias, both the participants and the recruitment research assistant will be blinded until allocation. The Result Research Assistant will not have access to the allocation base, nor to the allocation codes. On the other hand, it is declared that the intervention will be given by the researcher and that the main researcher will also participate in statistical analysis, therefore, the study is classified as single blind.

Measurement instruments

The information collection process will be carried out from the design of a form for the collection of sociodemographic data and clinical conditions of the participants and the application of the instruments for measuring both primary and secondary results:

* Self-management instrument in early stages CKD SM chronic kidney disease: 30 items, 4 factors (self-integration, problem solving, seeking social support and adherence to the recommended regimen), Cronbach's alpha of 0.95; English, Vietnamese, Taiwanese, and Mandarin languages. Likert scale evaluation, possible score from 29 to 116.
* Therapeutic adherence scale EAT: 21 items, 3 factors (control over the intake of drugs and food, medical-behavioral monitoring, and self-efficacy); Cronbach's alpha of 0.92, evaluation on a scale from 0 to 100; Spanish language.
* General Self-efficacy Scale: 10 items, Cronbach's alpha of 0.87, in English and Spanish languages.

MATERIALS AND METHODS

3.8.1 Study phases: for the satisfactory development of the study, the following phases will be found and carried out:

- Pre-pilot phase: In this phase, the following will be carried out: the adaptation of the CKD SMS intervention to the Colombian context, considering the evaluation by experts in the management of people with CKD in early stages (nephrologists, nephrology nurses, nutritionists, psychologists), the educational material of the intervention will be designed and created, which is also expected to be evaluated by experts.

On the other hand, in this phase, psychometric tests will be carried out to complete the validation of the instruments in the Colombian context, especially in the Self-Management instrument for people with CKD in early stages, which does not have a version in Spanish, where It will be carried out following the process as follows: It is proposed to carry out the cultural validation with semantic, linguistic and cultural analysis, translation and back translation, the content validity will be evaluated through a panel or expert judgment, based on the recommendations given by Tristan, following the following steps: 1. Define the objective and purpose of the expert judgment. 2. Selection of judges; minimum 5 considering academic training, experience, and recognition of the area. 3. Explain both the dimensions and the indicators that each of the items on the scale is measuring to assess whether it is indispensable, useful, and necessary. 4. Specify the purpose of the test. 5. Template design. 6. Calculate the agreement between judges by means of the content validity index. 7. Preparation of the conclusions of the trial. And for the construct validity, it will be done through exploratory and verifiable factor analysis; the reliability of the instrument will be made by means of Cronbach's alpha.

* Pilot Phase: In this phase, the field exploration will be carried out, followed by adjustments regarding the application time in the handling of the instruments and the training in these aspects for the research assistant, in addition to the intervention training for its implementation. optimal by the researcher.
* Main study phase - Recruitment of participants:

For the recruitment of participants, the following process will be carried out: 1. The database provided by the institution will be reviewed to identify the patients who can participate in the study, after which the randomization will be carried out. 2. The dates assigned for their control in the institution will be reviewed based on the chosen ones. 3. On the day of the consultation, the patient will be contacted and the information regarding the study will be presented, and if the participant shows interest in participating in it, the informed consent will be signed, and the instruments will be delivered to collect the data. baseline, before being assigned to the control or experimental group. 4. After the completion of the instruments, the patient will be given an envelope to choose for their random assignment, which contains a code, said code will be entered in a matrix, in which the main researcher can review who was assigned to the group experimental. 5. The main researcher, after verification of the codes assigned on the day, will contact each participant assigned to the experimental group to arrange the time to meet and start the intervention. 6. In a subsequent period of 16 weeks after entering the study, we will have contact with the participants from both the control group and the experimental group and the instruments will be applied again to obtain the data for the comparison of the effect.

This process will be carried out on the days when the nephrology consultation is carried out until the total number of participants calculated and assigned to each group is completed.

To report the flow of participants throughout the investigation, the CONSORT diagram for each group will be considered.

APPROACH TO THE ANALYSIS FRAMEWORK To respond to specific objectives 1 and 2, a statistical analysis will be carried out through descriptive statistics. Subsequently, a normality test will be carried out, to identify how the data distribution is presented, in addition, it is carried out to determine the tests to be used, whether parametric or non-parametric in the inferential analysis, bivariate and multivariate analysis. A bivariate analysis, to compare the sociodemographic and clinical characteristics between the groups.

To respond to specific objective 3, Inferential statistics will be carried out, which will be carried out to accept or reject the null or alternative hypothesis, which are proposed as:

* H1: The CKD SMS intervention in self-management in people with CKD in early stages is effective on self-management behaviors, self-efficacy, and therapeutic adherence. (H1: G1> G2; p <0.05)
* H0: The CKD SMS intervention in people with CKD in early stages is not effective on self-management behaviors, self-efficacy, and therapeutic adherence. (H0: G1 = G2; p> 0.05) But it is also used multivariate analysis, to determine the individual relationship but also the relationship of the possible variables that intervene on the results, a simple logistic regression model will be built and adjusted according to the possible confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Adults, of legal age for Colombia (18 years), with a diagnosis of chronic kidney disease in stages 1-4, without renal replacement therapy according to the Kdigo guidelines.
* People without comorbidity and with non-decompensated or exacerbated chronic comorbidities.
* People in use of their mental and communication faculties.

Exclusion Criteria:

* People who are under the effect of some substance that alters the mental state.
* People under 18 years of age.
* Being receiving renal replacement therapy or being in a terminal stage.
* Illiterate people.
* People who are participating in another educational intervention different from the usual care.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
self management | 4 month
  Self-management behaviors will be measured using the chronic kidney disease self-management instrument (CKD-SM), whose validity and reliability will be evaluated in the pre-pilot phase. The CKD-SM self-report instrument consists of 32 items and measures whether participants perform a variety of self-management behavior factors, including: self-integration (11 items); problem solving (11 items); search for social support (5 items); and adherence to the recommended regimen (5 items). The subscales are evaluated by adding the scores for each item using a Likert scale from 1 to 4; 1 = never, 2 = sometimes, 3 = usually, 4 = always. Total CKD-SM scores are also measured by summing the scores on the four subscales and can range from 32 to 128. High scores indicate a high level of CKD self-management behaviors

SECONDARY OUTCOMES:
Self-efficacy | 4 month
  Participants' self-efficacy will be measured using the general self-efficacy scale. Developed by Schwarzer and Jerusalem in 1995, composed of 10 items that are valued through a four-point Likert scale (1 = incorrect, 2 = hardly true, 3 = rather true, 4 = true). Higher scores indicate higher levels of self-efficacy
Therapeutic adherence | 4 month
  Therapeutic adherence will be measured by using the therapeutic adherence scale developed by Soria based on explicit behaviors, which includes information related to the therapeutic regimen, the interaction with health personnel, and self-efficacy to determine if the patient is able or not to be involved in the treatment. It contains 21 items evaluated with a scale from 0 to 100, subdivided into percentage ranges, of the self-reported type, where the score closer to 100 means that the person is more adherent

CONTACTS AND LOCATIONS:
Locations (1):
- Judith Medellin Olaya, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting in January 2025
Access Criteria: The information shared will be made through the database built with the information collected from the study where only the patients are identified by assigned codes to ensure their privacy, this information will only be shared with the study researchers, and will be shared in publications only information resulting from statistical analysis.

REFERENCES:
- [Background] Martinez-Castelao A, Gorriz JL, Segura-de la Morena J, Cebollada J, Escalada J, Esmatjes E, Facila L, Gamarra J, Gracia S, Hernand-Moreno J, Llisterri-Caro JL, Mazon P, Montanes R, Morales-Olivas F, Munoz-Torres M, de Pablos-Velasco P, de Santiago A, Sanchez-Celaya M, Suarez C, Tranche S. Consensus document for the detection and management of chronic kidney disease. Nefrologia. 2014;34(2):243-62. doi: 10.3265/Nefrologia.pre2014.Feb.12455. English, Spanish. PMID 24658201
- [Background] León-Hernándeza RC, Peñarrieta-de Córdovab M, Gutiérrez-Gómez T, Banda-Gonzálezd O, Flores-Barriose F, Rivera M. Self-management behavior predictors among persons with chronic diseases in Tamaulipas. Enfermería Univ [Internet]. 2019 [cited 2019 Sep 29];16(2):128-37. Available from: http://reddeautomanejo.com/assets/predictores-unam-2019.pdf
- [Background] Lewis RA, Lunney M, Chong C, Tonelli M. Identifying Mobile Applications Aimed at Self-Management in People With Chronic Kidney Disease. Can J Kidney Health Dis. 2019 Mar 13;6:2054358119834283. doi: 10.1177/2054358119834283. eCollection 2019. PMID 30899533
- [Background] Zimbudzi E, Lo C, Misso M, Ranasinha S, Zoungas S. Effectiveness of management models for facilitating self-management and patient outcomes in adults with diabetes and chronic kidney disease. Syst Rev. 2015 Jun 10;4:81. doi: 10.1186/s13643-015-0072-9. PMID 26059649
- [Background] Bonner A, Havas K, Douglas C, Thepha T, Bennett P, Clark R. Self-management programmes in stages 1-4 chronic kidney disease: a literature review. J Ren Care. 2014 Sep;40(3):194-204. doi: 10.1111/jorc.12058. Epub 2014 Mar 14. PMID 24628848
- [Background] Lee MC, Wu SV, Hsieh NC, Tsai JM. Self-Management Programs on eGFR, Depression, and Quality of Life among Patients with Chronic Kidney Disease: A Meta-Analysis. Asian Nurs Res (Korean Soc Nurs Sci). 2016 Dec;10(4):255-262. doi: 10.1016/j.anr.2016.04.002. Epub 2016 May 13. PMID 28057311
- [Background] Lin CC, Hwang SJ. Patient-Centered Self-Management in Patients with Chronic Kidney Disease: Challenges and Implications. Int J Environ Res Public Health. 2020 Dec 16;17(24):9443. doi: 10.3390/ijerph17249443. PMID 33339300
- [Background] Havas K, Douglas C, Bonner A. Person-centred care in chronic kidney disease: a cross-sectional study of patients' desires for self-management support. BMC Nephrol. 2017 Jan 13;18(1):17. doi: 10.1186/s12882-016-0416-2. PMID 28086812
- [Background] Gorostidi M, Santamaria R, Alcazar R, Fernandez-Fresnedo G, Galceran JM, Goicoechea M, Oliveras A, Portoles J, Rubio E, Segura J, Aranda P, de Francisco AL, Del Pino MD, Fernandez-Vega F, Gorriz JL, Luno J, Marin R, Martinez I, Martinez-Castelao A, Orte LM, Quereda C, Rodriguez-Perez JC, Rodriguez M, Ruilope LM. Spanish Society of Nephrology document on KDIGO guidelines for the assessment and treatment of chronic kidney disease. Nefrologia. 2014 May 21;34(3):302-16. doi: 10.3265/Nefrologia.pre2014.Feb.12464. Epub 2014 Mar 6. English, Spanish. PMID 24798565
- [Background] Lopez-Vargas PA, Tong A, Howell M, Craig JC. Educational Interventions for Patients With CKD: A Systematic Review. Am J Kidney Dis. 2016 Sep;68(3):353-70. doi: 10.1053/j.ajkd.2016.01.022. Epub 2016 Mar 26. PMID 27020884
- [Background] Havas K, Bonner A, Douglas C. Self-management support for people with chronic kidney disease: Patient perspectives. J Ren Care. 2016 Mar;42(1):7-14. doi: 10.1111/jorc.12140. Epub 2015 Sep 24. PMID 26404772
- [Background] Donald M, Kahlon BK, Beanlands H, Straus S, Ronksley P, Herrington G, Tong A, Grill A, Waldvogel B, Large CA, Large CL, Harwood L, Novak M, James MT, Elliott M, Fernandez N, Brimble S, Samuel S, Hemmelgarn BR. Self-management interventions for adults with chronic kidney disease: a scoping review. BMJ Open. 2018 Mar 22;8(3):e019814. doi: 10.1136/bmjopen-2017-019814. PMID 29567848
- [Background] Peñarrieta MI, Flores-Barrios F, Gutiérrez-Gómez T, Piñones -Martínez S, Resendiz -Gonzalez E, María Quintero-Valle L. Self-management and family support in chronic diseases. J Nurs Educ Pract [Internet]. 2015 [cited 2019 Oct 1];5(11). Available from: www.sciedu.ca/jnepURL:http://dx.doi.org/10.5430/jnep.vXnXpXX
- [Background] Lin MY, Liu MF, Hsu LF, Tsai PS. Effects of self-management on chronic kidney disease: A meta-analysis. Int J Nurs Stud. 2017 Sep;74:128-137. doi: 10.1016/j.ijnurstu.2017.06.008. Epub 2017 Jun 21. PMID 28689160
- [Background] Zimbudzi E, Lo C, Misso ML, Ranasinha S, Kerr PG, Teede HJ, Zoungas S. Effectiveness of self-management support interventions for people with comorbid diabetes and chronic kidney disease: a systematic review and meta-analysis. Syst Rev. 2018 Jun 13;7(1):84. doi: 10.1186/s13643-018-0748-z. PMID 29898785
- [Background] Nguyen NT, Douglas C, Bonner A. Effectiveness of self-management programme in people with chronic kidney disease: A pragmatic randomized controlled trial. J Adv Nurs. 2019 Mar;75(3):652-664. doi: 10.1111/jan.13924. Epub 2019 Feb 14. PMID 30537153
- [Background] Havas K, Douglas C, Bonner A. Meeting patients where they are: improving outcomes in early chronic kidney disease with tailored self-management support (the CKD-SMS study). BMC Nephrol. 2018 Oct 20;19(1):279. doi: 10.1186/s12882-018-1075-2. PMID 30342487
- [Background] Lin CC, Tsai FM, Lin HS, Hwang SJ, Chen HC. Effects of a self-management program on patients with early-stage chronic kidney disease: a pilot study. Appl Nurs Res. 2013 Aug;26(3):151-6. doi: 10.1016/j.apnr.2013.01.002. Epub 2013 Mar 7. PMID 23465757
- [Background] Peng S, He J, Huang J, Lun L, Zeng J, Zeng S, Zhang L, Liu X, Wu Y. Self-management interventions for chronic kidney disease: a systematic review and meta-analysis. BMC Nephrol. 2019 Apr 26;20(1):142. doi: 10.1186/s12882-019-1309-y. PMID 31027481
- [Background] Sorait W. The association of self-efficacy and self-management behavior in adult patients with chronic kidney disease: an integrative review. J Kidney Treat Diagnosis [Internet]. 2018 Jun 17 [cited 2020 Jul 4];1(1). Available from: https://www.pulsus.com/scholarly-articles/the-association-of-selfefficacy-and-selfmanagement-behavior-in-adult-patients-with-chronic-kidney-disease-an-integrative-review-4587.html
- [Background] Tung HH, Lien RY, Wei J, Clinciu DL, Lee JY, Huang HC. The role of adherence in the relationship between self-efficacy and self-management in diabetic patients undergoing CABG in Taiwan. Heart Asia. 2012 Sep 17;4(1):114-9. doi: 10.1136/heartasia-2012-010155. eCollection 2012. PMID 27326045

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05707260/Prot_SAP_000.pdf